CLINICAL TRIAL: NCT05736835
Title: A Phase 2 Trial of the Immunogenicity and Safety of CVXGA Intranasal COVID Vaccine in Healthy Adults
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CyanVac LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVXGA-002
Record Dates: First submitted 2023-02-17; First posted 2023-02-21 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: COVID-19
Keywords: COVID-19; intranasal vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CVXGA (Experimental): CVXGA single intranasal dose 10e7 PFU
  Interventions: Biological: CVXGA
- Placebo (Placebo Comparator): 0.9% sterile saline
  Interventions: Biological: CVXGA

INTERVENTIONS:
Biological: CVXGA — CVXGA is a live viral vector, consisting of a recombinant parainfluenza virus type 5 that carries the SARS-CoV-2 S-protein from WA.1 (not enrolling) or XBB1.5 strain.
  Other Names: PIV5-SARS CoV-2

SUMMARY:
The purpose of this trial is to evaluate immunogenicity and safety of CVXGA administered as a single intranasal dose against SARS-CoV-2 S-protein in participants. The trial will enroll up to 400 healthy participants, age 18-80 years.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, blinded study to evaluate the immunogenicity and safety of CVXGA.

Trial Population: Up to 400 healthy adults (18-80 years) that may have had prior COVID vaccination or COVID infection at least 5 months prior to planned study vaccine receipt.

Vaccine: CVXGA is a recombinant parainfluenza virus type 5 (PIV5) that carries the SARS-CoV-2 S protein. The vaccine will be administered as a single intranasal dose as a spray.

Study visits: Participants will be asked to complete 3 clinic visits and 1 follow-up phone call.

Participants >= 65 yrs of age will have an additional 2 clinic visits to test for vaccine shedding.

Follow-up will be for 6 months after single vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals ≥ 18 years and ≤ 80 years of age at the time of consent
2. Willing and able to comply with all scheduled visits, vaccination plan, laboratory tests and other study procedures
3. Determined by medical history, targeted physical examination and clinical judgement of the investigator to be in stable state of health. Screening laboratory values slightly outside lab normal ranges may be acceptable if the site investigator determines that they are not clinically significant.
4. Women of childbearing potential* must agree to use or have practiced true abstinence** or use at least one acceptable primary form of contraception.***, **** Note: These criteria are applicable to females in a heterosexual relationship and child-bearing potential (i.e., the criteria do not apply to subjects in a same sex relationship).*Not of childbearing potential: post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure® placement).**True abstinence is no sexual intercourse 100% of the time (i.e. male's penis never enters the female's vagina). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post- ovulation methods) and withdrawal are not acceptable methods of contraception.***Acceptable forms of primary contraception include monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the subject's vaccination, intrauterine devices, birth control pills, and injectable/implantable/insertable hormonal birth control products, condom, or diaphragm with spermicide. If barrier methods are to be used, then double barrier methods of protection are required, i.e., male condom, in combination with a cap, diaphragm, or sponge with spermicide.

   ****Must use at least one acceptable primary form of contraception for at least 28 days prior to vaccination and at least one acceptable primary form of contraception for 90 days after last vaccination. If barrier methods are to be used, then double barrier methods of protection are required, i.e., male condom, in combination with a cap, diaphragm, or sponge with spermicide.
5. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to each vaccination.
6. Male subjects of childbearing potential* must use condoms to ensure effective contraception with a female partner of childbearing potential from vaccination until 90 days after vaccination. Such female partners must also use an acceptable form of primary contraception as described under inclusion criterion #4. If barrier methods are to be used, then double barrier methods of protection are required, i.e., male condom, in combination with a cap, diaphragm, or sponge with spermicide.*Biological males who are post-pubertal and considered fertile until permanently sterile by bilateral orchiectomy or vasectomy.
7. Male subjects agree to refrain from sperm donation from the time of vaccination until 90 days after vaccination.
8. Female subjects agree to refrain from egg donation from time of vaccination until 90 days after vaccination.

Exclusion Criteria:

1. Receipt of approved or authorized COVID vaccine < 150 days prior to planned study vaccine administration or planned receipt of COVID vaccine during 6 months following receipt of study vaccine.
2. Covid infection (Positive COVID-19 test) < 150 days prior to planned study vaccine administration
3. Pregnant or breastfeeding participants.
4. History of severe COVID-19 infection (e.g., need for oxygenation or ventilatory support)
5. Receipt of SARS-CoV-2 immunoglobulin, monoclonal antibody or plasma antibody therapy < 150 days prior to study vaccine administration
6. Any prior receipt of a PIV5-based vaccine (e.g., CVXGA1 or BLB-201 [an RSV vaccine being developed by Blue Lake Biotechnology]).
7. Chronic rhinitis, nasal septal defect causing significant breathing problems, cleft palate, nasal polyps, or other nasal abnormality that might affect vaccine administration.
8. Current or planned simultaneous participation in another interventional study or receipt of any investigational study product within 28 days prior to study vaccine administration
9. A history of anaphylaxis, urticaria, or other significant adverse reaction requiring medical intervention after receipt of a vaccine (licensed or unlicensed).
10. A history of myocarditis or pericarditis at any time prior to enrollment, history of Kawasaki disease, or history of multisystem inflammatory syndrome after COVID infection.
11. Received or plans to receive a vaccine within 14 days prior to or after study vaccine.
12. Bleeding disorder diagnosed by a healthcare provider (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or bleeding difficulties with intramuscular injections or blood draws.
13. Current or previous diagnosis of a significant immunocompromising condition or other immunosuppressive condition.
14. Resides with someone who is severely immunocompromised.
15. Advanced liver or kidney diseases.
16. Advanced (CD4 count < 200) and/or untreated HIV, active Hepatitis B virus infection, positive serology for Hepatitis C.
17. Received oral, intramuscular or intravenous systemic immunosuppressants, or immune-modifying drugs for >14 days in total within 6 months prior to administration of study vaccine (for corticosteroids > / = 20 mg/day of prednisone equivalent).
18. History of significant/severe wheeze, respiratory symptoms resulting in hospitalization, or known bronchial hyperreactivity to viruses.
19. Received immunoglobulin or blood-derived products, within 3 months prior to study vaccine dose.
20. Received chemotherapy, immunotherapy or radiation therapy within 6 months prior to study vaccine dose.
21. Study personnel or an immediate family member or household member of study personnel.
22. Is acutely ill or febrile 72 hours prior to or at vaccine dosing day (fever defined as > / = 38.0 degrees Celsius /100.4 degrees Fahrenheit). Participants meeting this criterion may be rescheduled within the relevant window periods.
23. Receipt or anticipated receipt of, within 7 days prior to through 28 days after trial vaccination, any intranasal medication including FDA-approved prescription or over-the-counter products or non-FDA-approved alternative medicine products (e.g., Ayurvedic oil or other naturopathic substances).
24. Currently smoking or vaping, or history of regular smoking or vaping in the past two years
25. Active alcohol use disorder or alcohol abuse or active illicit drug abuse
26. Anticipated use of nasal irrigation (e.g., Neti Pot™) after enrollment through 28 days after trial vaccination.
27. Diagnosis of dementia or other cognitive deficit that might impact a participant's ability to understand the clinical trial or be compliant with trial procedures.
28. Planned hospital admission (e.g., for surgical or other invasive procedures) during the 6 months after trial enrollment that could interfere with study trial visits.
29. Planned admission or stay at an assisted living or other care facility during the 6 months after trial enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety outcome measures (SAEs, AEs, and local and systemic reactogenicity) | day 1-8, day 1-29, and day 1-181 post vaccination
  Percentage of subjects overall reporting:
  Local reactions for up to 7 days following vaccination (Day 1-8); Systemic events for up to 7 days following vaccination (Day 1-8); Adverse events (AEs) from Day 1 to 29; Serious AEs from Day 1 to 181; AESI from day 1 to 181; Comparison of the percentage of subjects reporting the events listed above compared with percentage of subjects in the placebo group
Immunogenicity | day 15 and day 29
  Proportion of subjects with an increase in GMFR from baseline for serum SARS-CoV-2 S-specific IgG and IgA antibodies (by ELISA) and/or an increase in SARS-CoV-2 S-protein specific cell mediated immune responses (CMI) in PBMC at Day 15 and/or Day 29 from baseline compared to proportion of placebo subjects.

SECONDARY OUTCOMES:
Secondary Safety | day 1 to 6 months
  Percentage of subjects reporting MAAEs or NOCMCs from Day 1 to 181 in CVXGA versus placebo group.
Secondary Immunogenicity | day 15 and day 29
  Proportion of subjects with an increase in nasal SARS-CoV-2 S-specific IgA at Day 15 and/or Day 29 from baseline compared to proportion of placebo subject

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jin, Study Chair — CyanVac LLC
Locations (10):
- United States (10):
  - Velocity Clinical Research, San Diego, California
  - Velocity Clinical Research, Boise, Idaho
  - Velocity Clinical Research, Sioux City, Iowa
  - Velocity Clinical Research, Rockville, Maryland
  - Velocity Clinical Research, Omaha, Nebraska
  - University of Rochester, Rochester, New York
  - Velocity Clinical Research, Vestal, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Velocity Clinical Research, Providence, Rhode Island
  - Velocity Clinical Research, Cedar Park, Texas

IPD SHARING:
Plan to Share IPD: No